CLINICAL TRIAL: NCT01326182
Title: Intervention for Depressed Latina Mothers of Children With Asthma
Acronym: MAADRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Elizabeth L. McQuaid, Prinicpal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4040-09; R21HL095102-01A1 (NIH)
Record Dates: First submitted 2010-07-08; First posted 2011-03-30 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2010-07

CONDITIONS: Pediatric Asthma; Maternal Depression
Keywords: asthma; depression; Latino
MeSH Terms: conditions — Asthma; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAADRE (Experimental): Group-based intervention combining asthma education and cognitive behavioral treatment for depressive symptoms
  Interventions: Behavioral: MAADRE
- MAAS (Active Comparator): Group-based treatment combining asthma education and general information regarding child health
  Interventions: Behavioral: MAAS

INTERVENTIONS:
Behavioral: MAADRE — Group-based intervention combining asthma education and CBT for depressive symptoms
  Arms: MAADRE
Behavioral: MAAS — Group-based intervention including asthma education and education regarding general child health
  Arms: MAAS

SUMMARY:
This study is to develop and pilot test a new group-based intervention for depressed Latina mothers of children with asthma. The investigators ongoing work has identified that close to 50% of Latina mothers of children with asthma report significant symptoms of depression. The intervention will combine asthma education and cognitive-behavioral strategies (e.g., increasing the pleasant activities that you do to help your mood) to address symptoms of depression. The investigators hope to improve mothers' mood, their feelings of confidence that they can manage asthma, and children's level of asthma control.

The project has two phases. In Phase 1, the investigators will develop the intervention by working on the treatment manual and then conducting focus groups with Latina mothers to get input on the intervention. The investigators expect 24 mothers at each of 2 sites (RI and PR) to participate in focus groups (8 mothers per group). The group will take approximately 1-1.5 hours.

In Phase 2, the investigators will conduct a small pilot of the intervention at both sites with new participants. At each site, 4 groups (4 sessions each) will be run. Participants will have an equal chance of being placed in the new intervention condition (asthma education and mood management), or in a control condition that covers asthma education and general topics regarding child health and wellness (e.g., encouraging reading, reducing screen time, nutrition). Participants will participate in a baseline research session, in the 4 intervention group sessions, and then in two follow-up research sessions (one at end of treatment which is expected to occur two months after enrollment, and one at 4-months post-treatment). They will complete survey instruments that assess their own depressive symptoms, family demographic characteristics, access/barriers to health care, self-efficacy to manage asthma, social network support, and family climate, as well as their child's asthma symptom frequency. Children 7-12 are included only for the assessment of asthma symptoms and lung function, which occurs at baseline, end of treatment, and 4-month follow up for 2 weeks at each time point. Participation in Phase 2 is expected to take approximately 6 months.

DETAILED DESCRIPTION:
Pediatric asthma, the most common childhood chronic illness, remains a significant public health problem. Research indicates marked health care disparities in asthma, with Latino children at particular risk for poor health outcomes. Maternal depressive symptoms are also high among poor women who have children with asthma, and may compromise effective asthma management. The first AIM of this R21 application is to develop a manualized treatment to integrate asthma education with CBT strategies to reduce depressive symptoms among Latina mothers of children with persistent asthma. Such an intervention has the potential to improve asthma outcomes through increasing maternal knowledge and self-efficacy to manage asthma. During Year 1, Expert Consultants and an investigator team with expertise in asthma education, culturally tailored treatment, and CBT for Latinos will provide input into the development of the integrated intervention (MAADRE, for its acronym in Spanish). Focus groups will be conducted with our target population in Rhode Island and Puerto Rico to refine intervention content. Qualitative data analyses will be used to prioritize intervention targets and to identify contextual differences between Island and Mainland groups. The second AIM of this application is to conduct a small two-site pilot of the MAADRE intervention in Rhode Island and Puerto Rico. During Year 2, the investigators will test the intervention with depressed mothers of children with asthma (32 in Puerto Rico and 32 in Rhode Island.) Mothers will be randomly assigned to receive either the MAADRE intervention or asthma education + child health (control). The investigators expect that target children of participants in the MAADRE intervention will have improved asthma outcomes (asthma symptom days, lung function as measured by FEV1 and FEV1/FVC, asthma-related quality of life, and asthma control) relative to the control condition. The investigators also anticipate that participants in the MAADRE intervention will have greater reduction in depressive symptoms and improved self-efficacy to manage asthma relative to the control condition. Findings from the proposed application will be used to design a larger RCT to evaluate the effects of the MAADRE intervention on asthma outcomes, and to compare cost-effectiveness of the intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

* Latina mothers with symptoms of depression and children with persistent asthma
* Ages 7-12 years old

Exclusion Criteria:

* serious suicidal risk
* significant psychopathology (psychosis)
* ethnicity other than Latino

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control | 2 months after baseline (end of treatment), 4 months post treatment
  Changes in Asthma Control from baseline will be assessed using the ACT at End of Treatment and 4 months post treatment

SECONDARY OUTCOMES:
Maternal Depression | 2 months after baseline (end of treatment), 4 months post treatment
  Changes in Maternal Depressive Symptoms from baseline will be evaluated using the Beck Depression Inventory at end of treatment and 4 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L McQuaid, PhD, Principal Investigator — Rhode Island Hospital
Locations (2):
- Rhode Island Hospital, Providence, Rhode Island, United States
- University of Puerto Rico, Rio Piedras, Puerto Rico